CLINICAL TRIAL: NCT03935672
Title: PEARL: PET-based Adaptive Radiotherapy Clinical Trial
Brief Title: PEARL PET-based Adaptive Radiotherapy Clinical Trial
Acronym: PEARL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Velindre NHS Trust (Other Government)
Responsible Party: Principal Investigator, Lisette Nixon, Senior Trial Manager, Velindre NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/VCC/0029; 242633 (Other: IRAS number)
Record Dates: First submitted 2018-10-03; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Oropharyngeal Cancer
Keywords: Oropharyngeal Cancer; Radiotherapy; HPV positive; Automated segmentation; Radiotherapy re-planning
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: PEARL is a prospective, interventional, non-randomised, phase II feasibility study for patients with good prognosis Human Papillomavirus (HPV)-associated oropharyngeal squamous cell cancer (OPSCC) who are suitable for treatment with concurrent chemo-radiotherapy (CCRT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All trial participants (Other): Baseline plasma and saliva tests for future translational analysis
  Baseline planning FDG PET CT scan
  Patients will start their 6 weeks of CCRT within two to three weeks following the planning scans. Cisplatin chemotherapy will be administered. 33 daily fractions of radiotherapy will be delivered over 6 weeks.
  A second FDG-PET-CT scan (iPET) and repeat plasma and saliva tests will be carried out after 2 weeks of CCRT (on RT days 9 - 12) and the iPET assessed for residual FDG-avid disease. The biological GTV will be re-outlined based on the residual avid region of the tumour on the second PET-CT (bGTV_iP)
  At the end of treatment, plasma and saliva tests will be carried out at 4 weeks post treatment and again at the 3 month post-treatment PET-CT
  Swallowing and QoL assessments will be repeated 4 weeks (+/- 2 weeks) after treatment and will be repeated at 6, 12 and 24 months post-treatment. The plasma and saliva samples will be repeated at 12 and 24 months
  Interventions: Procedure: PET-CT scans; Procedure: Outlining the biological GTVs (bGTV_P and bGTV_iP); Procedure: Blood samples for cell-free DNA analysis; Procedure: Salivary samples for cell-free DNA analysis

INTERVENTIONS:
Procedure: PET-CT scans — Patients will have three scans during the trial.
  * The 1st scan (prePET) is a baseline diagnostic scan. The patient is in a thermoplastic shell and PET CT will be used by to define a bGTV_P. bGTV_P will then be used as an adjunct to help us delineate the GTV_P.
  * The 2nd scan (iPET) takes place following 2 weeks (10 fractions) of chemo-radiotherapy. The patient is in a thermoplastic shell and the PET CT will be used to delineate the remaining avid disease (bGTV_iP).
  * The 3rd scan takes place 3 months following the last dose of radiotherapy. It will be used to ascertain whether any avid disease remains and may inform the need for further treatment.
Procedure: Outlining the biological GTVs (bGTV_P and bGTV_iP) — The biological GTVs (bGTV_P and bGTV_iP) will be automatically delineated by ATLAAS and verified manually by a nuclear medicine physician and a clinical oncologist. It will consist of the high FDG uptake volume based on visual assessment whilst using suitable windowing levels. Any differences in contouring will be settled either by the two doctors reaching a consensus or by a third doctor if differences between the first two cannot be resolved.
Procedure: Blood samples for cell-free DNA analysis — In order to contribute to our understanding of how disease processes may be monitored in a less invasive and less morbid manner, we will be collecting blood and saliva samples prior to, during, and after the radical treatment of OPSCC in PEARL, to see if there is correlation with disease status and FDG-PET-CT response.
Procedure: Salivary samples for cell-free DNA analysis — In order to contribute to our understanding of how disease processes may be monitored in a less invasive and less morbid manner, we will be collecting blood and saliva samples prior to, during, and after the radical treatment of OPSCC in PEARL, to see if there is correlation with disease status and FDG-PET-CT response.

SUMMARY:
The PEARL study will recruit approximately 50 patients with human papillomavirus (HPV)-positive oropharyngeal squamous cell carcinoma (OPSCC) who are about to undergo primary treatment with concurrent chemo-radiation from South Wales (Velindre Cancer Centre and Singleton Hospital, Swansea) and Bristol. The main aim is to see whether it is feasible to preform a positron emission tomography-computed tomography (PET-CT) scan after 2 weeks of radiotherapy and re-plan the radiotherapy based on this PET-CT scan, to re-distribute the dose of radiotherapy being delivered, so that a smaller area of normal tissues in the mouth and throat are treated to a high dose of radiotherapy.

DETAILED DESCRIPTION:
PEARL is a prospective, interventional, non-randomised, phase II feasibility study for patients with good prognosis Human Papillomavirus (HPV)-associated oropharyngeal squamous cell cancer (OPSCC) who are suitable for treatment with concurrent chemo-radiotherapy (CCRT).

The incidence of oropharyngeal squamous cell carcinoma (OPSCC) caused by Human Papillomavirus (HPV) infection (HPV-positive OPSCC) is increasing in the United Kingdom. It tends to affect younger patients and has a better outcome than most other head and neck cancers.

A large proportion of patients diagnosed with HPV-positive OPSCC will undergo non-surgical treatment. This usually involves 6 to 7 weeks of chemo-radiotherapy, with chemotherapy being given weekly or during the first and fourth week of the radiotherapy course (CCRT). Many patients with HPV-positive OPSCC are cured of their disease but often have to live for several decades with the side effects of their treatment. Side effects from radiotherapy are usually caused because normal tissues surrounding the cancer receive radiation whilst the cancer itself is being treated.

Positron emission tomography-computed tomography (PET-CT) scans are able to look at the metabolic (or biological) activity of cells and are currently recommended in the UK for response assessment after a patient has completed radiotherapy for a head and neck cancer but, as far as we know, have not yet been used routinely to adapt radiotherapy according to the individual patient's response during radiotherapy.

PEARL will explore the feasibility of individually adapting the radiotherapy plan for each patient after 2 weeks of radical CCRT, based on biological changes in tumour activity seen on an interim FDG-PET-CT scan, carried out early on during a course of treatment. The aim is to reduce the dose of radiotherapy received by surrounding normal tissues to ultimately reduce toxicity.

The study will establish the progression free survival rate (PFS) in patients who receive biologically adapted radiotherapy. Furthermore, it will also explore whether changes seen on PET-CT scan during treatment correlate with outcome and with changes in potential blood-based biomarkers of response. Toxicity rates will be assessed, particularly the effect of treatment on swallowing function.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the oropharynx
2. Positive p16 Immunohistochemistry on local testing
3. UICC TNM (8th edition) stage T1 - T3 N0 - N1 M0
4. Multidisciplinary team (MDT) decision to treat with primary chemoradiotherapy
5. Patients considered fit for radical treatment with primary chemoradiotherapy (including sufficient renal function (GFR>50ml/min)
6. Aged 18 years or older
7. Not smoked in the last 2 years
8. Written informed consent provided
9. Patients with reproductive potential (male or female), who are sexually active during the duration of the trial consent to using a highly effective method of contraception for at least six months after the last dose of chemoradiotherapy. Effective forms of contraception are described in section 15.5.

Exclusion Criteria:

1. Known HPV negative squamous cell carcinoma of the head and neck
2. T1 - T3 tumours where primary treatment with concomitant chemo-radiotherapy is not considered appropriate
3. T4 disease
4. N2 (TMN8) nodal disease
5. Distant metastatic disease
6. Current smokers or smokers who have stopped within the past 2 years
7. Diabetes mellitus
8. Any pre-existing medical condition likely to impair swallowing function and/ or a history of pre-existing swallowing dysfunction prior to index oropharyngeal cancer
9. Previous radiotherapy to the head and neck
10. History of malignancy in the last 5 years, except basal cell carcinoma of the skin, or carcinoma in situ of the cervix
11. Tumour non-avid on PET-CT or not visible on cross sectional imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression free survival at 2 years | 2 years following enrolment
  To maintain a high progression free survival rate with biologically adapted radiotherapy in patients with good prognosis HPV positive OPSCC. To be certain that we are not having a negative impact on PFS by adapting the RT plan we will ensure that PFS is at least as high as expected after treatment with chemo-radiotherapy in patients with similarly staged HPV-positive OPSCC.

SECONDARY OUTCOMES:
Monthly recruitment rate | End of 2 years recruitment period
  As this is a feasibility study, recruitment will be monitored and monthly recruitment rate over 2 years will be presented.
To test if individualized, adaptive, biologically-based radiotherapy planning is feasible and results in a significant change in the radiotherapy plan. | 2 weeks (10 fractions) of chemo-radiotherapy
  Percentage reduction in mean dose to OAR (superior pharyngeal constrictor muscles, contralateral parotids, contralateral submandibular gland, salivary glands) as a result of PET-CT during treatment. Percentage change to PTV will also be presented.
To test if individualized, adaptive, biologically-based radiotherapy planning results in a significant change in the radiotherapy plan. | 2 weeks (10 fractions) of chemo-radiotherapy
  Percentage reduction in mean dose to OAR (superior pharyngeal constrictor muscles, contralateral parotids, contralateral submandibular gland, salivary glands) as a result of PET-CT during treatment. Percentage change to PTV will also be presented.
To maintain high complete response rates 3 months after treatment | 3 months post treatment
  The proportion of patients who are complete metabolic responders at 3 months as per PERCIST criteria will be presented.
Acute toxicity rates | 3 months post treatment
  Cumulative acute CTCAE toxicity score percentages during and up to 3 months after treatment will be presented.
Late toxicity rates | 6, 12 and 24 months post treatment
  Water swallow test will be plotted over time, scores will be presented at 6, 12, 18 and 24 months.
Late toxicity rates | 6, 12 and 24 months post treatment]
  MDADI will be plotted over time, scores will be presented at 6, 12, 18 and 24 months.
Late toxicity rates | 6, 12 and 24 months post treatment]
  QoL scores will be plotted over time, scores will be presented at 6, 12, 18 and 24 months.
To assess the effect of treatment on swallowing function | 3, 6, 12 and 24 months post treatment
  Water swallow test scores will be plotted over time.
To assess the effect of treatment on swallowing function | 3, 6, 12 and 24 months post treatment
  MDADI scores will be plotted over time.
To assess the effect of treatment on swallowing function | 3, 6, 12 and 24 months post treatment
  QoL scores will be plotted over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mererid Evans, Principal Investigator — Velindre Cancer Centre
Locations (3):
- United Kingdom (3):
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Singleton Hospital, Swansea, Wales
  - University Hospitals Bristol NHS Foundation Trust, Bristol

IPD SHARING:
Plan to Share IPD: Undecided